CLINICAL TRIAL: NCT00235495
Title: A Phase III Randomized Multicenter Clinical Trial Of High-Dose Human Albumin Therapy For Neuroprotection In Acute Ischemic Stroke
Brief Title: Albumin in Acute Ischemic Stroke Trial
Acronym: ALIAS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment halted by DSMB following interim analysis.
Sponsor: University of Miami (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Calgary (Other); Medical University of South Carolina (Other); Neurological Emergencies Treatment Trials Network (NETT) (Network)
Responsible Party: Principal Investigator, Myron Ginsberg, Principal Investigator; Peritz Scheinberg Professor of Neurology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20060083; U01NS054630 (NIH); NIH NINDS 5U01 NS040406-08 (Other: Internal tracking number); 20060233 (Other: Western IRB)
Record Dates: First submitted 2005-09-14; First posted 2005-10-10 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Ischemic Stroke
Keywords: stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Albumins; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albumin (ALB) (Active Comparator): Albumin (human albumin, 25% solution, 2.0 g/kg), infused intravenously over a period of 2 hours
  Interventions: Biological: Albumin
- Saline (Placebo Comparator): Saline (isotonic solution), 8 ml/kg, infused intravenously over a 2-hour period
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: Albumin — human albumin, 25%, 2.0g/kg intravenously (or equivalent volume of saline control), infused over 2 h, commencing within 5 hours of stroke onset
  Arms: Albumin (ALB)
Drug: Saline — equivalent volume of isotonic saline control
  Arms: Saline

SUMMARY:
The goal of the trial is to determine whether human albumin, administered within 5 hours of symptom onset, improves the 3-month outcome of subjects with acute ischemic stroke.

DETAILED DESCRIPTION:
Human serum albumin, at 2 g/kg, administered over 2 hours by intravenous infusion, will be compared to placebo (isovolumic normal saline) among patients with acute ischemic stroke. All patients will have a baseline stroke severity measured as NIH Stroke scale score > 5. Patients will treated according to the best standard of care including concurrent treatment with intravenous or intra-arterial thrombolysis where appropriate. The primary outcome will be determined at 3 months. The primary hypothesis is that, using the composite outcome of a modified Rankin score 0-1 or NIH stroke scale score 0-1 at 3 months (or both), the proportion of patients with improved outcomes will be greater by 10% or more in the active treatment group. [The current trial is termed "Part 2" and incorporates revisions to the initial protocol that were instituted after the Data Safety Monitoring Board (DSMB) suspended subject recruitment because of a safety concern after 434 subjects had been enrolled. The protocol revisions of Part 2 resulted from the study team's thorough review of the Part-1 safety data and were designed to optimize safety going forward.]

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke
* NIH stroke scale score > 5
* Age >= 18 and <= 83
* ALB or placebo can be administered within 5 hours of symptom onset
* ALB or placebo can be administered within 60 minutes of Tissue Plasminogen Activator (tPA) administration in the thrombolysis group
* Signed informed consent

Exclusion Criteria:

* Episode/exacerbation of congestive heart failure (CHF) from any cause in the last 6 months. An episode of congestive heart failure is any heart failure that required a change in medication, diet or hospitalization.
* Known valvular heart disease with CHF in the last 6 months.
* Severe aortic stenosis or mitral stenosis.
* Cardiac surgery involving thoracotomy (e.g., coronary artery bypass graft (CABG), valve replacement surgery) in the last 6 months.
* Acute myocardial infarction in the last 6 months.
* Signs or symptoms of acute myocardial infarction, including ECG findings, on admission.
* Baseline elevated serum troponin level on admission (>0.1 mcg/L)
* Suspicion of aortic dissection on admission.
* Acute arrhythmia (including any tachycardia - or bradycardia) with hemodynamic instability.
* Findings on physical examination of any of the following: (1) jugular venous distention (JVP > 4 cm above the sternal angle); (2) 3rd heart sound; (3) resting tachycardia (heart rate > 100/min) attributable to congestive heart failure; (4) abnormal hepatojugular reflux; (5) lower extremity pitting edema attributable to congestive heart failure; and/or (6) definite chest x-ray evidence of pulmonary edema.
* Current acute or chronic lung disease requiring supplemental chronic or intermittent oxygen therapy.
* Historical Modified Rankin Score (mRS) ≥2. Patients who live in a nursing home or who are not fully independent for activities of daily living immediately prior to the stroke are not eligible for the trial.
* In-patient stroke. I.e., patients with a stroke occurring as a complication of hospitalization for another condition, or as a complication of a procedure.
* Planned acute use of intra-arterial (IA) tPA or acute endovascular intervention (e.g., stenting, angioplasty, thrombus retrieval device use) must conform to the following criteria: (1) begin within 5 hours of symptom onset, and (2) finish within 7 hours of symptom-onset.
* Fever, defined as core body temperature > 37.5° C (99.5°F).
* Serum creatinine > 2.0 mg/dL or 180 µmol/L.
* Profound dehydration.
* Evidence of intracranial hemorrhage (intracerebral hematoma (ICH), subarachnoid hemorrhage (SAH), epidural hemorrhage, acute or chronic subdural hematoma (SDH)) on the baseline CT or MRI scan.
* History of allergy to albumin.
* History of latex rubber allergy.
* Severe chronic anemia with Hgb < 7.5 g/dL
* Pregnancy, breastfeeding or positive pregnancy test. (Women of childbearing age must have a negative pregnancy test prior to ALB administration.)
* Concurrent participation in any other therapeutic clinical trial.
* Evidence of any other major life-threatening or serious medical condition that would prevent completion of 3-month follow-up, impair the assessment of outcome, or in which ALB therapy would be contraindicated or might cause harm to the subject.

Ages: 18 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 841 (Actual)
Dates: Start 2006-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron D. Ginsberg, MD, Study Chair — University of Miami; Michael D. Hill, MD MSc, Principal Investigator — University of Calgary; Yuko Y Palesch, PhD, Principal Investigator — Medical University of South Carolina
Locations (89):
- United States (69):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - University of Arizona Medical Center-South Campus, Tucson, Arizona
  - University of Arizona Medical Center, Tucson, Arizona
  - John Muir Medical Ctr-Concord, Concord, California
  - El Camino Hospital, Mountain View, California
  - UCSF Medical Center, San Francisco, California
  - UCSF-San Francisco General Hospital, San Francisco, California
  - California Pacific Medical Center, Davies Campus, San Francisco, California
  - California Pacific Medical Center, Pacific Campus, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - UCLA Medical Center, Santa Monica, Santa Monica, California
  - Stanford University Medical Center, Stanford, California
  - John Muir Medical Ctr-Walnut Creek, Walnut Creek, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Christiana Hospital, Newark, Delaware
  - University of Florida/Shands, Jacksonville, Florida
  - Jackson Memorial Hospital, University of Miami, Miami, Florida
  - The Villages Research Group, Ocala, Florida
  - Neuroscience Research Institute at Florida Hospital Orlando, Orlando, Florida
  - Intercoastal Neurology/Medical Research Center, Sarasota, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - St. Elizabeth Medical Center South, Edgewood, Kentucky
  - St. Elizabeth Hospital, Florence, Kentucky
  - University of Kentucky Hospital, Lexington, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Upper Chesapeake Medical Center, Bel Air, Maryland
  - Detroit Receiving Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Sinai-Grace Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Fairview Southdale Hospital, Edina, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - HealthEast Care System/St. Joseph's Hospital, Saint Paul, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Atlantic Neuroscience Institute, Overlook Hospital, Summit, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Buffalo General Medical Center, Buffalo, New York
  - Mercy Hospital of Buffalo, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Med Health and Hospitals, Raleigh, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Mercy Health Fairfield Hospital, Fairfield, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - OHSU Legacy Emmanuel Hospital, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Sacred Heart Medical Center, Springfield, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Seton Medical Center, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Froedtert Memorial Hospital, Milwaukee, Wisconsin
- Canada (13):
  - Foothills Hospital, University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Royal Island Hospital, Kamloops, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia
  - London Health Sciences Centre-University Hospital, London, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - University of Toronto, St. Michael's Hospital, Toronto, Ontario
  - Hopital Charles LeMoyne, Centre de Recherche, Greenfield Park, Quebec
  - Centre de Sante et de Service Sociaux de Chicoutimi, Saguenay, Quebec
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Tampere University Hospital, Tampere
- Israel (5):
  - Hadassah Medical Organization, Hadassah University Hospital, ‘En Kerem, Jerusalem
  - Chaim Sheba Medical Center at Tel-Hashomer, Tel Litwinsky, Ramat Gan
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Tel-Aviv Sourasky Medical Center, Tel Aviv

REFERENCES:
- [Derived] Martin RH, Yeatts SD, Hill MD, Moy CS, Ginsberg MD, Palesch YY; ALIAS Parts 1 and 2 and NETT Investigators. ALIAS (Albumin in Acute Ischemic Stroke) Trials: Analysis of the Combined Data From Parts 1 and 2. Stroke. 2016 Sep;47(9):2355-9. doi: 10.1161/STROKEAHA.116.012825. Epub 2016 Jul 26. PMID 27462118
- [Derived] Hill MD, Martin RH, Palesch YY, Moy CS, Tamariz D, Ryckborst KJ, Jones EB, Weisman D, Pettigrew C, Ginsberg MD. Albumin Administration in Acute Ischemic Stroke: Safety Analysis of the ALIAS Part 2 Multicenter Trial. PLoS One. 2015 Sep 1;10(9):e0131390. doi: 10.1371/journal.pone.0131390. eCollection 2015. PMID 26325387
- [Derived] Ginsberg MD, Palesch YY, Hill MD, Martin RH, Moy CS, Barsan WG, Waldman BD, Tamariz D, Ryckborst KJ; ALIAS and Neurological Emergencies Treatment Trials (NETT) Investigators. High-dose albumin treatment for acute ischaemic stroke (ALIAS) Part 2: a randomised, double-blind, phase 3, placebo-controlled trial. Lancet Neurol. 2013 Nov;12(11):1049-58. doi: 10.1016/S1474-4422(13)70223-0. Epub 2013 Sep 27. PMID 24076337
- [Derived] Hill MD, Martin RH, Palesch YY, Tamariz D, Waldman BD, Ryckborst KJ, Moy CS, Barsan WG, Ginsberg MD; ALIAS Investigators; Neurological Emergencies Treatment Trials Network. The Albumin in Acute Stroke Part 1 Trial: an exploratory efficacy analysis. Stroke. 2011 Jun;42(6):1621-5. doi: 10.1161/STROKEAHA.110.610980. Epub 2011 May 5. PMID 21546491

RESULTS

PARTICIPANT FLOW:
Groups:
- Albumin: Treatment with 25% Albumin, 2.0 g/kg
- Saline: Treatment with same volume of normal saline
Period: Overall Study
Arm/Group | Albumin | Saline
Started | 422 | 419
Completed | 354 | 351
Not Completed | 68 | 68
Not completed — Death | 52 | 42
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Lost to Follow-up | 11 | 13
Not completed — Visit/assessmen outside window/missing | 0 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Albumin | Saline | Total
Number analyzed (Participants) | 422 | 419 | 841
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 202 | 188 | 390
  >=65 years | 219 | 231 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.42 (12.95) | 64.84 (12.88) | 64.13 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 184 | 386
  Male | 220 | 235 | 455
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 26 | 50
  Not Hispanic or Latino | 379 | 372 | 751
  Unknown or Not Reported | 19 | 21 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native/First Nations People | 2 | 0 | 2
  Asian | 25 | 20 | 45
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black | 69 | 86 | 155
  White | 314 | 305 | 619
  Multiple, Other, or Unknown | 10 | 7 | 17
Oxfordshire Community Stroke Project Classification [Count of Participants; unit: Participants]
  Total Anterior Circulation Syndrome | 102 | 98 | 200
  Partial Anterior Circulation Syndrome | 232 | 235 | 467
  Posterior Circulation Syndrome | 35 | 39 | 74
  Lacunar Stroke | 53 | 47 | 100
Baseline National Institutes of Health Stroke Scale (NIHSS) Score [Median (Inter-Quartile Range); unit: units on a scale] — The National Institutes of Health Stroke Scale (NIHSS) is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. The scores range from 0 to 42 with a score of greater than 20 indicating severe neurologic deficit.
  units on a scale | 11 [8 to 17] | 11 [8 to 17] | 11 [8 to 17]
Baseline ASPECTS [Number; unit: Participants]
  Baseline ASPECTS >7 | 325 | 327 | 652
  Baseline ASPECTS <= 7 | 93 | 88 | 181
  Missing | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Favorable Outcome Defined as National Institute of Health Stroke Scale (NIHSS) Score of 0-1 and/or Modified Rankin Scale (mRS) of 0-1.
Description: The National Institutes of Health Stroke Scale (NIHSS) is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. The scores range from 0 to 42 with a score of greater than 20 indicating severe neurologic deficit. The mRS ranges from 0-6 representing perfect health without symptoms to death. A score of 0 is no symptoms at all and a score of 1 is no significant disability. Able to carry out all usual duties and activities.
Time Frame: at 3 months
Population: Intent to Treat population - All subjects randomized into the study are included and analyzed based on the treatment arm to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 422 | 419
Participants | 186 | 185
Statistical Analysis 1: Comparison: Albumin vs Saline; Test of null hypothesis (equal proportions of subjects with NIHSS 0-1 or mRS 0-1 or both at 90 days post-randomization in Albumin and Saline treatment arms) versus alternative hypothesis (greater proportion of subjects with NIHSS 0-1 or mRS 0-1 or both at 90 days post-randomization in Albumin treatment arm); Test type: Superiority or Other; Regression, Logistic — The generalized linear model with log link function is tested at the one-sided alpha level of 0.025; Adjustment is made for baseline NIHSS and Thrombolysis stratum; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.84 to 1.10] — Adjusted risk ratio greater than 1 indicates greater risk of good outcome in the Albumin treatment group, while adjusted risk ratio less than 1 indicates greater risk of good outcome in the Saline treatment group

2. Secondary Outcome: Number of Participants With a Composite Outcome of mRS 0-1 and/or NIHSS 0-1 and/or Decrease in NIHSS From Baseline by 10 or More Points
Time Frame: at 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 422 | 419
Participants | 227 | 241
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 0.93, 99% CI 2-sided [0.80 to 1.09]

3. Secondary Outcome: Number of Participants With a NIHSS of 0-1 at 24 Hours
Description: The National Institutes of Health Stroke Scale (NIHSS) is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. The scores range from 0 to 42 with a score of greater than 20 indicating severe neurologic deficit.
Time Frame: at 24 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 422 | 419
Participants | 65 | 62
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 0.99, 99% CI 2-sided [0.66 to 1.49]

4. Secondary Outcome: Number of Participants With a NIHSS 0-1 at 90 Days.
Description: as for outcome 3
Time Frame: at 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 422 | 419
Participants | 65 | 62
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 0.88, 99% CI 2-sided [0.71 to 1.10]

5. Secondary Outcome: The Number of Participants With a Score on the mRS 0-1 at 90 Days.
Description: The mRS ranges from 0-6 representing perfect health without symptoms to death. 0 = No symptoms at all. 1 = No significant disability. Able to carry out all usual duties and activities. 2 = Slight disability. Unable to carry out all previous activities but able to look after own affairs without assistance. 3 = Moderate disability. Requires some help, but able to walk unassisted. 4 = Moderately severe disability. Unable to walk unassisted and unable to attend to own bodily needs without assistance. 5 = Severe disability. Bedridden, incontinent, and requires constant nursing care and attention. 6 = Dead.
Time Frame: at 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 422 | 419
Participants | 155 | 145
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 1.03, 99% CI 2-sided [0.82 to 1.28]

6. Secondary Outcome: The Number of Participants With a Score on the mRS of 0-2 at 90 Days.
Description: as for outcome 5
Time Frame: at 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 422 | 419
Participants | 227 | 221
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 0.99, 99% CI 2-sided [0.85 to 1.13]

7. Secondary Outcome: Number of Participants With a Favorable Outcome Per Modified Rankin Scare (mRS)
Description: Assessed as the final global disability level on the modified Rankin scale (mRS) at 90 days better than expectation (sliding dichotomy analysis) ) assessed in the intention to treat population.
  mRS Scale:
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 422 | 419
Participants | 142 | 141
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 0.98, 99% CI 2-sided [0.87 to 1.11]

8. Secondary Outcome: Barthel Index (BI) 95-100
Description: The Barthel Index (BI) is an ordinal scale used to measure a subject's performance in activities of daily living (ADL) in ten variables - feeding, transfer (bed to chair), grooming, toilet use, bathing, mobility on a level surface, stair use, dressing, bowels and bladder. It is an assessment of independence in ADL and is scored in increments of 5 points. the highest total score for fully independent subjects equals 100. A higher number is associated with a greater likelihood of being able to live at home with a degree of independence.
Time Frame: at 90 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 422 | 419
participants
  BI 95-100 | 227 | 231
  Otherwise | 195 | 188
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 0.95, 99% CI 2-sided [0.83 to 1.10]

9. Secondary Outcome: Number of Participants With an EuroQol (EQ-5D) Favorable Score < 0.78
Description: The EQ-5D measures the subject's overall health state in a descriptive system of health-related quality of life (QoL) states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which can take one of three responses. The responses record three levels of severity ('no problems', 'some problems', and 'extreme problems) within a particular EQ-5D dimension. The EQ-5D results can be converted to health utility scores.
Time Frame: at 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 422 | 419
Participants | 155 | 152
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 0.99, 99% CI 2-sided [0.84 to 1.17]

10. Secondary Outcome: Number of Participants With a Stroke Specific Quality of Life Scale (SSQOL) Score of >=3
Description: Stroke, specific, health-related quality of life (SSQoL) is a self-reported survey that includes 12 domains and 49 items which are scored on a 5pt Likert response format with a lower score indicating worse function/lower ability on that item or domain. Domain scores were calculated as an unweighted average of item scores in that domain. Overall Total Score was calculated as an unweighted average of domain scores. Each Domain Score and the Overall Total Score all range from 1-5 with 1 being worst and 5 being the best. We have presented data here for the number of participants that have an unweighted average of domain scores of 3 or greater.
Time Frame: at 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 422 | 419
Participants | 258 | 268
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 0.93, 99% CI 2-sided [0.84 to 1.02]

11. Secondary Outcome: Trailmaking A
Description: The Trail Making Test is a neuropsychological test of visual attention and task switching that is thought to be sensitive to the presence of cerebral dysfunction. It is a timed test consisting of two parts where the subject is asked to draw a "trail" made by connecting numbers in sequential order (part A) and then in part B the combination of numbers and letters. Scoring is calculated separately for Parts A and B but both scores are provided as the minutes and seconds it takes for the subject to complete ach part. Normally, the entire test (A and B) can be completed in 5-10 minutes.
Time Frame: at 90 days
Population: Participants were excluded if the Tail Making Test was not assessed.
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 269 | 272
Minutes | 55 [39 to 105] | 56 [39 to 90]
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; p = 0.913, Wilcoxon rank sum test, normal approx; Rank Sum = 73098

12. Secondary Outcome: Trailmaking B
Description: as for outcome 11
Time Frame: at 90 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 215 | 210
Minutes | 111 [78 to 173] | 110 [82 to 180]
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; p = 0.923, Wilcoxon rank sum test, normal approx; Rank Sum = 44853.5

13. Secondary Outcome: Number of Participants With Neurological Deterioration Within 48 Hours
Description: This is assessed as the number of participants with a neurological adverse event.
Time Frame: within 48 hours
Population: The safety sample consisted of the 830 subjects who received at least 20% of the indented dose of study-drug. In order to be considered for this analysis, subject must have had the event within the time frame or been followed for at least 48 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 411 | 412
Participants | 47 | 40
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 1.18, 95% CI 2-sided [0.79 to 1.76]

14. Secondary Outcome: Neurological Death Within 7 Days
Time Frame: within 7 days
Population: The safety sample consisted of the 830 subjects who received at least 20% of the indented dose of study-drug. In order to be considered for this analysis, subject must have had the event within the time frame or been followed for at least 7 days.
Measure: Number; unit: participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 404 | 407
participants | 13 | 13
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.47 to 2.15]

15. Secondary Outcome: Recurrent Ischemic Stroke Within 30 Days
Time Frame: within 30 days
Population: The safety sample consisted of the 830 subjects who received at least 20% of the indented dose of study-drug. In order to be considered for this analysis, subject must have had the event within the time frame or been followed for at least 30 days.
Measure: Number; unit: participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 373 | 370
participants | 7 | 6
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 1.16, 95% CI 2-sided [0.39 to 3.41]

16. Secondary Outcome: Atrial Fibrillation Within 48 Hours
Time Frame: within 48 hours
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 410 | 412
participants | 32 | 19
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 1.69, 95% CI 2-sided [0.98 to 2.94]

17. Secondary Outcome: Pulmonary Edema Within 48 Hours
Time Frame: within 48 hours
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 412 | 412
participants | 54 | 5
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 10.8, 95% CI 2-sided [4.37 to 26.72]

18. Secondary Outcome: Shortness of Breath Within 48 Hours
Time Frame: within 48 hours
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 410 | 412
participants | 18 | 7
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 2.58, 95% CI 2-sided [1.09 to 6.12]

19. Secondary Outcome: Symptomatic Intracerebral Hemorrhage (ICH) Within 24 Hours
Time Frame: within 24 hours
Population: The safety sample consisted of the 830 subjects who received at least 20% of the indented dose of study-drug. In order to be considered for this analysis, subject must have had the event within the time frame or been followed for at least 24 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 415 | 414
Participants | 17 | 7
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 2.42, 95% CI 2-sided [1.02 to 5.78]

20. Secondary Outcome: Asymptomatic ICH Within 24 Hours
Time Frame: within 24 hours
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 415 | 414
Participants | 27 | 23
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 1.14, 95% CI 2-sided [0.68 to 2.01]

21. Secondary Outcome: Death Within 30 Days
Time Frame: within 30 days
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 409 | 406
participants | 39 | 37
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.68 to 1.61]

22. Secondary Outcome: Death Within 90 Days
Time Frame: within 90 days
Population: The safety sample consisted of the 830 subjects who received at least 20% of the indented dose of study-drug. In order to be considered for this analysis, subject must have had the event within the time frame or been followed for at least 90 days.
Measure: Number; unit: participants
Arm/Group | Albumin | Saline
Number analyzed (Participants) | 378 | 369
participants | 46 | 41
Statistical Analysis 1: Comparison: Albumin vs Saline; Test type: Superiority or Other; Regression, Logistic; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.74 to 1.63]

ADVERSE EVENTS:
Arm/Group | Albumin | Saline
Serious Adverse Events (participants affected / at risk) | 212/422 | 178/419
Other Adverse Events (participants affected / at risk) | 352/422 | 341/419
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albumin (N=422) | Saline (N=419)
FEVER (General disorders) | 1 (1) | 2 (2)
BACTEREMIA (Infections and infestations) | 0 (0) | 1 (1)
SEPTICEMIA OR SEPTIC SHOCK (Infections and infestations) | 3 (3) | 5 (6)
OROLINGUAL ANGIOEDEMA (Immune system disorders) | 2 (2) | 2 (2)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
LOCALIZED PAIN (General disorders) | 1 (1) | 1 (1)
SYSTEMIC HEMORRHAGE (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
FAILURE TO THRIVE (General disorders) | 3 (3) | 1 (1)
OTHER SYSTEMIC ADVERSE EVENT OR COMPLICATION (General disorders) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 22 (26) | 12 (13)
ACUTE RESPIRATORY DISTRESS SYNDROME (ARDS) OR RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4)
PULMONARY EMBOLISM (Vascular disorders) | 7 (7) | 5 (5)
APNEA OR RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY INSUFFICIENCY (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER RESPIRATORY DISORDER OR COMPLICATION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
ANGINA PECTORIS (STABLE) (Cardiac disorders) | 1 (1) | 1 (1)
ACUTE CORONARY SYNDROME - MYOCARDIAL INFARCTION (Cardiac disorders) | 13 (15) | 9 (9)
CARDIAC ARREST (Cardiac disorders) | 2 (2) | 6 (6)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 0 (0)
"CONGESTIVE HEART FAILURE, PULMONARY EDEMA" (Cardiac disorders) | 21 (21) | 6 (7)
PERIPHERAL ARTERIAL OCCLUSION (Cardiac disorders) | 1 (1) | 0 (0)
VENTRICULAR FIBRILLATION OR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION/FLUTTER (Cardiac disorders) | 10 (11) | 3 (3)
BRADYCARDIA (Cardiac disorders) | 3 (5) | 2 (2)
"CONDUCTION BLOCKS (ATRIO-VENTRICULAR BLOCKS, BUNDLE-BRANCH BLOCKS)" (Cardiac disorders) | 2 (2) | 0 (0)
SUPRAVENTRICULAR ARRHYTHMIAS (Cardiac disorders) | 0 (0) | 3 (3)
DEEP VENOUS THROMBOSIS (Cardiac disorders) | 1 (1) | 4 (4)
ARTERIAL DISSECTION (Cardiac disorders) | 0 (0) | 1 (1)
ARTERIAL EMBOLUS (Cardiac disorders) | 0 (0) | 1 (1)
HYPERTENSION-NOT INTENDED (Vascular disorders) | 1 (1) | 1 (1)
HYPOTENSION-NOT INTENDED (Vascular disorders) | 3 (3) | 5 (5)
ACUTE CORONARY SYNDROME - UNSTABLE ANGINA (Cardiac disorders) | 1 (1) | 0 (0)
CHEST PAIN (INCLUDING ATYPICAL) WITHOUT MENTION OF CARDIAC ORIGEN (Cardiac disorders) | 3 (3) | 4 (4)
TROPONIN LEAK (Cardiac disorders) | 1 (1) | 0 (0)
VALVULAR HEART DISEASE (Cardiac disorders) | 1 (1) | 1 (1)
PRE-CEREBRAL OR CEREBRAL VASCULAR DISEASE (INCLUDING STENOSIS OR OCCLUSION) (Vascular disorders) | 10 (10) | 8 (8)
OTHER CARDIAC ARRHYTHMIAS (Cardiac disorders) | 1 (1) | 2 (2)
OTHER CARDIOVASCULAR DISORDER OR COMPLICATION (Cardiac disorders) | 10 (10) | 13 (14)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTRIC OR DUODENAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA/VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL TRACT BLEEDING (Gastrointestinal disorders) | 7 (7) | 11 (12)
DYSPHAGIA (Gastrointestinal disorders) | 2 (2) | 0 (0)
PARALYTIC ILEUS/ BOWEL PSEUDO-OSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
BOWEL OSBTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER DIGESTIVE DISORDER OR COMPLICATION (Gastrointestinal disorders) | 7 (10) | 9 (10)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
OTHER ENDOCRINE OR METABOLIC DISORDER OR COMPLICATION (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
NON-CEREBRAL HEMORRHAGE (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
COAGULOPATHY (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
RECURRENT STROKE NOT SPECIFIED AS HEMORRHAGE OR INFARCTION (Nervous system disorders) | 16 (16) | 16 (19)
DEPRESSION OF CONSCIOUSNESS (Nervous system disorders) | 2 (2) | 0 (0)
BRAIN ABSCESS OR ENCEPHALITIS (Nervous system disorders) | 1 (1) | 0 (0)
MENINGITIS OR VENTRICULITIS (Nervous system disorders) | 0 (0) | 1 (1)
SYMPTOMATIC INTRACRANIAL HEMORRHAGE (Blood and lymphatic system disorders) | 22 (22) | 8 (8)
ASYMPTOMATIC INTRACRANIAL HEMORRHAGE (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
TRANSIENT ISCHEMIC ATTACK (Nervous system disorders) | 6 (8) | 10 (10)
CEREBRAL INFARCTION (Nervous system disorders) | 4 (4) | 12 (14)
CEREBRAL EDEMA (Nervous system disorders) | 16 (18) | 16 (16)
SEIZURE (Nervous system disorders) | 18 (23) | 15 (18)
CONFUSION/ENCEPHALOPATHY/DELIRIUM (Nervous system disorders) | 1 (1) | 1 (1)
ANXIETY (Nervous system disorders) | 3 (3) | 2 (2)
HEADACHE (Nervous system disorders) | 3 (3) | 6 (6)
INCREASED INTRA-CRANIAL PRESSURE (Nervous system disorders) | 1 (1) | 0 (0)
PROGRESSION OF STROKE (Nervous system disorders) | 15 (17) | 16 (17)
SYNCOPE OR PRE-SYNCOPE (Vascular disorders) | 4 (8) | 7 (7)
OTHER NEUROLOGICAL DISORDER OR COMPLICATION (Nervous system disorders) | 16 (17) | 13 (13)
URINARY TRACT INFECTION (Infections and infestations) | 5 (8) | 9 (9)
HEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL INSUFFICIENCY (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 2 (2) | 3 (3)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER UROGENITAL DISORDER OR COMPLICATION (Renal and urinary disorders) | 1 (1) | 5 (7)
FRACTURE (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
SURGICAL SITE INFECTION (Infections and infestations) | 4 (4) | 0 (0)
SURGICAL WOUND HEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER NON-INFECTIOUS SURGICAL WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
DECUBITUS ULCERS/PRESSURE SORES (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
MALIGNANT NEOPLASM (EXCEPT SKIN) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 8 (8)
PSYCHIATRIC DEPRESSION (Psychiatric disorders) | 2 (3) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
"HEMATOMA, NOT OTHERWISE SPECIFIED" (Vascular disorders) | 2 (2) | 1 (1)
PSYCHIATRIC DISORDER (Psychiatric disorders) | 4 (4) | 1 (3)
CELLULITIS/NON-SURGICAL SKIN INFECTION (Infections and infestations) | 2 (2) | 2 (2)
OTHER UNCLASSIFIED ADVERSE EVENT (General disorders) | 11 (12) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albumin (N=422) | Saline (N=419)
FEVER (General disorders) | 38 (42) | 34 (35)
BACTEREMIA (Infections and infestations) | 3 (3) | 2 (2)
SEPTICEMIA OR SEPTIC SHOCK (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
OROLINGUAL ANGIOEDEMA (Immune system disorders) | 1 (1) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 16 (16) | 14 (16)
ITCHING (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
ALLERGIC REACTION TO STUDY DRUG (Immune system disorders) | 3 (3) | 2 (2)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
LOCALIZED PAIN (General disorders) | 54 (73) | 55 (78)
GENERALIZED PAIN (General disorders) | 9 (10) | 9 (9)
CRAMPING (Reproductive system and breast disorders) | 7 (7) | 6 (7)
SYSTEMIC HEMORRHAGE (Blood and lymphatic system disorders) | 11 (12) | 11 (11)
FATIGUE (General disorders) | 2 (2) | 2 (2)
DIZZINESS (Nervous system disorders) | 6 (6) | 9 (9)
OTHER SYSTEMIC ADVERSE EVENT OR COMPLICATION (General disorders) | 17 (18) | 12 (12)
PNEUMONIA (Infections and infestations) | 31 (33) | 23 (25)
ACUTE RESPIRATORY DISTRESS SYNDROME (ARDS) OR RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
PULMONARY EMBOLISM (Vascular disorders) | 1 (1) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
HYPOXEMIA (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
HYPERCARBIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
CRACKLES/RALES (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (6)
APNEA OR RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
TACHYPNEA (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7)
RESPIRATORY INSUFFICIENCY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 7 (9)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 7 (7)
UPPER REPIRATORY INFECTION (Infections and infestations) | 9 (9) | 11 (11)
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 11 (11)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
OTHER RESPIRATORY DISORDER OR COMPLICATION (Respiratory, thoracic and mediastinal disorders) | 33 (45) | 36 (49)
ANGINA PECTORIS (STABLE) (Cardiac disorders) | 2 (2) | 2 (2)
ACUTE CORONARY SYNDROME - MYOCARDIAL INFARCTION (Cardiac disorders) | 4 (4) | 0 (0)
"CONGESTIVE HEART FAILURE, PULMONARY EDEMA" (Cardiac disorders) | 41 (45) | 14 (14)
VENTRICULAR FIBRILLATION OR TACHYCARDIA (Cardiac disorders) | 2 (2) | 3 (3)
ATRIAL FIBRILLATION/FLUTTER (Cardiac disorders) | 40 (42) | 35 (36)
BRADYCARDIA (Cardiac disorders) | 27 (27) | 32 (34)
TACHYCARDIA (Cardiac disorders) | 12 (14) | 17 (17)
"CONDUCTION BLOCKS (ATRIO-VENTRICULAR BLOCKS, BUNDLE-BRANCH BLOCKS)" (Cardiac disorders) | 4 (5) | 1 (1)
SUPRAVENTRICULAR ARRHYTHMIAS (Cardiac disorders) | 6 (8) | 1 (1)
DEEP VENOUS THROMBOSIS (Vascular disorders) | 6 (6) | 11 (12)
SUPERFICIAL VENOUS THROMBOSIS (Vascular disorders) | 2 (2) | 2 (2)
ARTERIAL DISSECTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ARTERIAL THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
HYPERTENSION-NOT INTENDED (Vascular disorders) | 39 (42) | 29 (31)
HYPOTENSION-NOT INTENDED (Vascular disorders) | 19 (21) | 33 (36)
CHEST PAIN (INCLUDING ATYPICAL) WITHOUT MENTION OF CARDIAC ORIGEN (Cardiac disorders) | 4 (4) | 13 (15)
TROPONIN LEAK (Cardiac disorders) | 51 (53) | 20 (20)
VALVULAR HEART DISEASE (Cardiac disorders) | 6 (8) | 8 (16)
EKG ABNORMALITIES (Investigations) | 8 (8) | 7 (7)
PHLEBITIS (Infections and infestations) | 1 (1) | 0 (0)
PRE-CEREBRAL OR CEREBRAL VASCULAR DISEASE (INCLUDING STENOSIS OR OCCLUSION) (Vascular disorders) | 6 (6) | 5 (5)
FLUID OVERLOAD ALONE (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
OTHER CARDIAC ARRHYTHMIAS (Cardiac disorders) | 12 (15) | 10 (13)
OTHER CARDIOVASCULAR DISORDER OR COMPLICATION (Cardiac disorders) | 23 (34) | 23 (31)
ABDOMINAL PAIN (Gastrointestinal disorders) | 13 (13) | 15 (15)
GASTRITIS/ ESOPHAGITIS/GERD (Gastrointestinal disorders) | 8 (8) | 7 (10)
GASTRIC OR DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 2 (2)
NAUSEA/VOMITING (Gastrointestinal disorders) | 70 (81) | 48 (54)
GASTROINTESTINAL TRACT BLEEDING (Gastrointestinal disorders) | 5 (5) | 7 (8)
"HEPATITIS, JAUNDICE, OR LIVER FAILURE" (Hepatobiliary disorders) | 0 (0) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 15 (15) | 9 (10)
CONSTIPATION (Gastrointestinal disorders) | 30 (34) | 48 (51)
FECAL INCONTINENCE (Gastrointestinal disorders) | 2 (2) | 2 (2)
LIVER ENZYMES ELEVATION (Investigations) | 6 (6) | 9 (9)
DYSPHAGIA (Gastrointestinal disorders) | 4 (4) | 2 (2)
PARALYTIC ILEUS/ BOWEL PSEUDO-OSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
BOWEL OSBTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER DIGESTIVE DISORDER OR COMPLICATION (Gastrointestinal disorders) | 33 (39) | 38 (49)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 34 (35) | 31 (31)
DIABETES INSIPIDUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 (2) | 6 (6)
HYPONATREMIA (Metabolism and nutrition disorders) | 5 (5) | 9 (9)
HYPERNATREMIA (Metabolism and nutrition disorders) | 11 (11) | 4 (4)
HYPOKALEMIA (Metabolism and nutrition disorders) | 93 (99) | 66 (72)
HYPERKALEMIA (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
HYPERLIPIDEMIA (Metabolism and nutrition disorders) | 8 (8) | 21 (21)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 6 (6) | 11 (11)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 18 (19) | 18 (18)
DEHYDRATION (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
ACID-BASE IMBALANCE (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
HYPOCHLOREMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
HYPERCHLOREMIA (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
OTHER ENDOCRINE OR METABOLIC DISORDER OR COMPLICATION (Metabolism and nutrition disorders) | 36 (47) | 42 (63)
NON-CEREBRAL HEMORRHAGE (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 16 (18) | 25 (29)
COAGULOPATHY (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
ANEMIA (Blood and lymphatic system disorders) | 39 (43) | 29 (34)
POLYCYTEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 15 (15) | 13 (14)
TROMBOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER COAGULATION OR HEMATOLOGIC DISORDER OR COMPLICATION (Blood and lymphatic system disorders) | 5 (5) | 8 (9)
RECURRENT STROKE NOT SPECIFIED AS HEMORRHAGE OR INFARCTION (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
DEPRESSION OF CONSCIOUSNESS (Nervous system disorders) | 10 (11) | 7 (7)
SYMPTOMATIC INTRACRANIAL HEMORRHAGE (Blood and lymphatic system disorders) | 7 (7) | 6 (6)
ASYMPTOMATIC INTRACRANIAL HEMORRHAGE (Blood and lymphatic system disorders) | 45 (48) | 35 (39)
CRANIAL NERVE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TRANSIENT ISCHEMIC ATTACK (Vascular disorders) | 2 (3) | 3 (3)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL EDEMA (Nervous system disorders) | 8 (10) | 10 (11)
SEIZURE (Nervous system disorders) | 10 (10) | 7 (9)
CONFUSION/ENCEPHALOPATHY/DELIRIUM (Psychiatric disorders) | 5 (5) | 6 (6)
ANXIETY (Psychiatric disorders) | 9 (9) | 12 (12)
HEADACHE (Nervous system disorders) | 81 (92) | 76 (84)
AGITATION (Nervous system disorders) | 15 (16) | 22 (24)
APHASIA (Psychiatric disorders) | 1 (2) | 1 (1)
INCREASED INTRA-CRANIAL PRESSURE (Nervous system disorders) | 1 (1) | 0 (0)
PROGRESSION OF STROKE (Nervous system disorders) | 18 (18) | 9 (9)
RETINAL VASCULAR ACCIDENT (Eye disorders) | 1 (1) | 0 (0)
SYNCOPE OR PRE-SYNCOPE (Vascular disorders) | 3 (3) | 3 (3)
OTHER NEUROLOGICAL DISORDER OR COMPLICATION (Nervous system disorders) | 31 (38) | 39 (46)
URINARY TRACT INFECTION (Infections and infestations) | 73 (81) | 72 (83)
HEMATURIA (Renal and urinary disorders) | 19 (19) | 18 (18)
RENAL INSUFFICIENCY (Renal and urinary disorders) | 11 (12) | 8 (9)
RENAL FAILURE (Renal and urinary disorders) | 2 (2) | 3 (3)
UROGENITAL INCONTINENCE (WAS 410) (Renal and urinary disorders) | 6 (6) | 5 (5)
URINARY RETENTION (Renal and urinary disorders) | 11 (13) | 12 (13)
OTHER UROGENITAL DISORDER OR COMPLICATION (Renal and urinary disorders) | 21 (23) | 25 (31)
FRACTURE (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
INFILTRATION OF IV SITE (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
SURGICAL SITE INFECTION (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
SURGICAL WOUND HEMATOMA (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
OTHER NON-INFECTIOUS SURGICAL WOUND COMPLICATION (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
DECUBITUS ULCERS/PRESSURE SORES (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (9)
BLISTER (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
MALIGNANT NEOPLASM (EXCEPT SKIN) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MALIGNANT NEOPLASM (SKIN) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ACCIDENTAL TRAUMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PSYCHIATRIC DEPRESSION (Psychiatric disorders) | 32 (34) | 35 (35)
FALL (Injury, poisoning and procedural complications) | 14 (15) | 13 (15)
PERIPHERAL EDEMA (General disorders) | 16 (19) | 16 (23)
OTHER ENZYME/S ELEVATION (Investigations) | 3 (3) | 2 (3)
INSOMNIA (Psychiatric disorders) | 19 (19) | 29 (30)
"HEMATOMA, NOT OTHERWISE SPECIFIED" (Vascular disorders) | 12 (12) | 8 (10)
DERMATITIS (Skin and subcutaneous tissue disorders) | 4 (5) | 6 (6)
PSYCHIATRIC DISORDER (Psychiatric disorders) | 2 (2) | 5 (5)
CELLULITIS/NON-SURGICAL SKIN INFECTION (Infections and infestations) | 14 (16) | 11 (14)
OTHER UNCLASSIFIED ADVERSE EVENT (General disorders) | 40 (49) | 40 (54)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No